CLINICAL TRIAL: NCT00331058
Title: A Study To Validate Key Therapeutic Targets and Characterise Their Response to Corticosteroids in Multiple Asthma Phenotypes
Brief Title: Comparison Of Molecular Targets In Mild To Severe Asthmatics And Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was truncated due to the long period of enrollment and the collection of a sufficient amount of data that allowed the scientific objectives to be met
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RES100767
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: Severe Asthma bronchoscopy
MeSH Terms: conditions — Asthma | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Other): control group not receiving prednisolone
  Interventions: Procedure: Prednisolone
- asthmatic volunteers (Other): receive prednisolone for 14-16 days
  Interventions: Procedure: Bronchoscopsy

INTERVENTIONS:
Procedure: Bronchoscopsy — Healthy and Asthmatic Volunteers
  Arms: asthmatic volunteers
Procedure: Prednisolone — Asthmatic Volunteers
  Arms: healthy volunteers

SUMMARY:
The primary goal of this study is to compare the expression of key GSK drug targets across the 4 asthma phenotypes and healthy subjects and secondarily to evaluate changes in target expression in response to a 2-week course of corticosteroids across the 4 asthma phenotypes. Each asthmatic subject in this study will undergo two bronchoscopies. Each healthy subject will undergo one bronchoscopy.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects aged between 18-60 years inclusive at screening.
* A female subject of childbearing potential must be using effective contraceptive
* measures described in protocol for at least one month prior to Screening and should continue using the same contraceptive measure during the study until completion of follow-up procedures. Non child-bearing potential is defined as pre-menopausal females with documented (medical report verification) hysterectomy or surgical sterilisation, or post-menopausal women who have been amenorrheic for more than 1 year and having estradiol and FSH levels consistent with menopause.). Other methods include male partner who is sterile prior to female subject's entry into study and is the sole sexual partner for that female subject.
* Atopic or non-atopic subjects
* Able to comprehend the nature of this research protocol and other relevant medical information and the ability to give written informed consent prior to participation in the study.
* Able to comply with the requirements and restrictions listed in the consent form.
* Available to complete the study and all measurements.
* Read, comprehend, and write English at a sufficient level to complete study related materials.

Additional inclusion criteria for the steroid naïve intermittent asthmatics - Cohort A

* Have a pre-history of a physician's diagnosis of asthma, with exclusion of other significant pulmonary
* No significant disease other than asthma.
* No history of steroid myopathy.
* No history of recent exposure to live vaccine in the past 4 weeks and no intention to undergo live vaccination during the prednisolone trial or during the month following the trial.
* Intermittent asthma with FEV1 ≥ 80% predicted.
* Positive beta agonist reversibility as shown by greater than 12% improvement on FEV1or greater than 200ml improvement in FEV1 within 30 minutes following the administration of Albuterol Inhalation Aerosol OR a positive PC20 to Methacholine Challenge smaller than 16 mcg.
* Not currently taking inhaled steroids (ICS), and has not taken ICS for at least 6 months prior to screening.
* A non-smoker (as demonstrated by a negative urine cotinine) for at least the past 12 months with a pack history ≤5 pack years.

Additional inclusion criteria for the mild to moderate persistent asthmatics on regular inhaled steroids - Cohort B

* Have a pre-history of a physician's diagnosis of asthma, with exclusion of other significant pulmonary diseases
* No significant disease other than asthma.
* No history of steroid myopathy.
* No history of recent exposure to live vaccine in the past 4 weeks and no intention to undergo live vaccination during the prednisolone trial or during the month following the trial.
* Mild to moderate persistent asthmatic with FEV1 ≥ 80% predicted
* Asthma symptoms ranging from daily to less than once a day
* Positive beta agonist reversibility as shown by greater than 12% improvement on FEV1or greater than 200ml improvement in FEV1 within 30 minutes following the administration of Albuterol Inhalation Aerosol OR a positive PC20 to Methacholine Challenge smaller than 16 mcg.
* On regular inhaled steroid treatment (from 200-500 mcg FP daily or equivalent). Short and long acting beta-2 agonists, anti-cholinergies, and Leukotriene receptor antagonists are allowed as concurrent medication.
* A non-smoker (as demonstrated by a negative urine cotinine) for at least the past 12 months with a pack history ≤5 pack years.

Additional inclusion criteria for the severe persistent asthmatics on maximal therapy; regular oral steroids - Cohort C

* Have a pre-history of a physician's diagnosis of asthma, with exclusion of other significant pulmonary diseases
* No significant disease other than asthma.
* No history of steroid myopathy.
* No history of recent exposure to live vaccine in the past 4 weeks and no intention to undergo live vaccination during the prednisolone trial or during the month following the trial.
* Severe persistent asthmatic
* Subjects should have at least one (if on oral steroids) or two (if only on inhaled steroids) of the following indices:

  1. FEV1 <80% (post bronchodilator) and FEV1/FVC ratio <70% predicted;
  2. Daily symptoms ± nocturnal symptoms as recorded in diary cards during run-in;
  3. severe exacerbations (as defined FACET study Tattersfield 1999) of ≥ twice a year in at least one of the last two years, as recorded in clinical records
* Positive beta agonist reversibility as shown by greater than 12% improvement on FEV1 or greater than 200ml improvement in FEV1 within 30 minutes following the administration of Albuterol Inhalation Aerosol OR a positive PC20 to Methacholine Challenge smaller than 16 mcg.
* High dose inhaled steroids (≥ to 1000 mcg FP daily or equivalent), oral steroids of ≤ 20mg prednisolone a day or equivalent.
* A non-smoker (as demonstrated by a negative urine cotinine) for at least the past 12 months with a pack history ≤5 pack years.

Additional inclusion criteria for the currently smoking, mild to moderate persistent asthmatics on maximal therapy; regular oral steroids - Cohort D

* Have a pre-history of a physician's diagnosis of asthma, with exclusion of other significant pulmonary
* No significant disease other than asthma.
* No history of steroid myopathy.
* No history of recent exposure to live vaccine in the past 4 weeks and no intention to undergo live vaccination during the prednisolone trial or during the month following the trial.
* Smokers (as demonstrated by a positive urine cotinine) with a pack history >5 pack years
* Mild to moderate persistent asthmatic with FEV1 ≥ 80% predicted
* Asthma symptoms less than once a day
* Positive beta agonist reversibility as shown by greater than 12% improvement on FEV1or greater than 200ml improvement in FEV1 within 30 minutes following the administration of Albuterol Inhalation Aerosol OR a positive PC20 to Methacholine Challenge smaller than 16mcg.
* On regular inhaled steroid treatment (200-500 mcg FP daily or equivalent). (NB:

short and long acting beta-2 agonists, anti-cholinergies, and Leukotriene receptor antagonists are allowed as concurrent medication.) Additional inclusion criteria for healthy volunteers, non asthmatic, non smokers - Cohort E Healthy; defined as individuals who are free of significant cardiovascular, pulmonary (e.g. tuberculosis), gastrointestinal, hepatic, endocrine, renal, haematological, neurological and psychiatric disease as determined by medical history, physical examination and clinical chemistry/haematology/urinalysis investigation.

• A non-smoker (as demonstrated by a negative urine cotinine) for at least the past 12 months with a pack history ≤5 pack years.

Exclusion criteria:

* As a result of medical interview, physical examination or screening investigation the physician responsible considers the subject unfit for the study.
* The subject has a history of drug or other allergy, which, in the opinion of the responsible physician, contra-indicates their participation.
* Subject is female who is pregnant or lactating.
* Having participated within 30 days or 5 half-lives in a study receiving an investigational drug.
* Having participated within 30 days in a study with an invasive procedure.
* Donation of a 500 mL of blood within the previous 56 days or intention to donate within 56 days of the end of the last bronchoscopy.
* Evidence of recent infection that would preclude participation in the steroid trial in the judgement of the study physician. The subject may be deferred to later participation. History of abnormal bruising or bleeding.
* History of alcohol or drug abuse within five years.
* Positive urine test for drugs of abuse including alcohol at screen.
* Abnormal (clinically significant) clinical laboratory test results.
* Medical history of cirrhosis, hepatitis C or hepatitis B or HIV
* Doing night-shift work that will change pattern within at least 5 days prior to study start through the first follow up visit for Cohorts A through D. This does not include the follow up visits at 6 and 12 months.
* Female subjects who are unwilling or unable to use an appropriate method of contraception
* Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
* Concomitant medications that may interfere with study procedures or evaluations.
* History of hypersensitivity to any of the following medications: Lidocaine, Fentanyl, Versed, Demerol, Midazolam, Epinephrine, Flumanzenil and Naloxon.
* History of hypersensitivity to bronchodilator (such as Albuterol)
* ALL WOMEN OF CHILD BEARING POTENTIAL WHO DO NOT WISH TO USE PROTOCOL APPROVED METHODS OF CONTRACEPTION WILL BE EXCLUDED.

Additional exclusion criteria for the steroid naïve intermittent asthmatics - Cohort A

* Subject has changed asthma medication within 1 month prior to screening.
* Subject had an asthma exacerbation in the previous month.
* Known sensitivity or allergy to prednisolone.
* History of tuberculosis, glaucoma, epilepsy, severe affective disorder or peptic ulceration.
* Current use or use within the previous 1 month of oral corticosteroids.
* Current use of any asthma medication except short acting inhaled β2 agonists
* Current use of Methotrexate, cyclosporin, PDE inhibitors, azathioprine or other immunosuppressive agents, except steroids.

Additional exclusion criteria for the mild to moderate persistent asthmatics on regular inhaled steroids - Cohort B

* Subject has changed asthma medication within 1 month prior to screening.
* Subject had an asthma exacerbation in the previous month.
* Known sensitivity or allergy to prednisolone.
* History of tuberculosis, glaucoma, epilepsy, severe affective disorder or peptic ulceration.
* Current use or use within the previous 1 month of oral corticosteroids.
* Current use of Methotrexate, cyclosporin, PDE inhibitors, azathioprine or other immunosuppressive agents, except steroids.

Additional exclusion criteria for the severe persistent asthmatics on maximal therapy; regular oral steroids - Cohort C

* Subject has changed asthma medication within 1 month prior to screening.
* Subject had an asthma exacerbation in the previous month.
* Known sensitivity or allergy to prednisolone.
* History of tuberculosis, glaucoma, epilepsy, severe affective disorder or peptic ulceration.
* Current use or use within the previous 1 month of oral prednisolone or equivalent of greater than 20mg daily.
* Current use of Methotrexate, cyclosporin, PDE inhibitors, azathioprine or other immunosuppressive agents, except steroids.
* Subjects should avoid any medications that in the opinion of the physician might interfere with either the safety of the subject or the interpretation of the results (e.g.

anti-inflammatory drugs)

Additional exclusion criteria for the currently smoking, mild to moderate persistent currently smoking asthmatics on regular inhaled steroids - Cohort D

* Subject has changed asthma medication within 1 month prior to screening.
* Subject had an asthma exacerbation in the previous month.
* Known sensitivity or allergy to prednisolone.
* History of tuberculosis, glaucoma, epilepsy, severe affective disorder or peptic ulceration.
* Current use or use within the previous 1 month of oral corticosteroids.
* Current use of Methotrexate, cyclosporin, PDE inhibitors, azathioprine or other immunosuppressive agents, except steroids.

Additional exclusion criteria for the healthy volunteers, non asthmatic non smokers - Cohort E The subject has any history of breathing problems in adult life (i.e. history of asthmatic symptoms). Screening lung function tests (FEV1) will be performed to confirm normal lung function parameters (≥80% predicted).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2006-02-18 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

PRIMARY OUTCOMES:
compare key drug targets across 4 asthma phenotypes and healthy subjects | visits 3 through to and including visit 6
evaluate changes in target expression in response to a 2 week course of corticosteroids across the 4 asthma phenotypes | visits 3 through to and including visit 6

SECONDARY OUTCOMES:
Histopathology on bronchial biopsies | visits 3 through to and including visit 6
Cytospins | visits 3 through to and including visit 6
target protein expression | visits 3 through to and including visit 6
target expression in the blood | visits 3 through to and including visit 6
inflammatory markers | visits 3 through to and including visit 6
lung function | visits 3 through to and including visit 6
Radiological Parameters | visits 3 through to and including visit 6
Quality of life (QoL) and symptom scores | visits 3 through to and including visit 6
Changes in medication | visits 3 through to and including visit 6
Measures of pulmonary inflammation | visits 3 through to and including visit 6
Assessments of lung structure | visits 3 through to and including visit 6
activation state of a signalling pathway | visits 3 through to and including visit 6
Whole Blood TaqMan and/or transcriptomic analysis | visits 3 through to and including visit 6
new targets and biomarkers | visits 3 through to and including visit 6
TaqMan and/or Differential Gene Expression and Proteomics | visits 3 through to and including visit 6
Pharmacogenomics from blood samples | visits 3 through to and including visit 6

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Siddiqui S, Shikotra A, Richardson M, Doran E, Choy D, Bell A, Austin CD, Eastham-Anderson J, Hargadon B, Arron JR, Wardlaw A, Brightling CE, Heaney LG, Bradding P. Airway pathological heterogeneity in asthma: Visualization of disease microclusters using topological data analysis. J Allergy Clin Immunol. 2018 Nov;142(5):1457-1468. doi: 10.1016/j.jaci.2017.12.982. Epub 2018 Mar 14. PMID 29550052
- See also: Results for study RES100767 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/RES100767?search=study&search_terms=RES100767#rs